CLINICAL TRIAL: NCT07201597
Title: Correlation Between Psychological Readiness, Knee Function and Isokinetic Performance After Anterior Cruciate Ligament Reconstruction
Brief Title: Correlation Between Psychological Readiness, Knee Function, and Isokinetic Performance After Anterior Cruciate Ligament Reconstruction (ACLR) Using Peroneus Longus Tendon Graft (PL-ACL-2025)
Acronym: PL-ACLR
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Al Hayah University In Cairo (Other)
Responsible Party: Principal Investigator, Mostafa Hamdy Abdelaziz Nagy, Demonstrator of Physical Therapy, Al Hayah University In Cairo
Other Study IDs: PL-ACL-2025
Record Dates: First submitted 2025-09-20; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament (ACL) Injury; Athletic Injuries; Knee Injuries
Keywords: ACL Injury; ACL Reconstruction; Peroneus Longus Tendon; Return to Sport; Psychological Readiness; Knee Function; Isokinetic Strength Testing; Hamstring-to-Quadriceps Ratio; Post-Surgery Rehabilitation; Sports Medicine; Physical Therapy Rehabilitation; Knee Stability; peroneus longus graft
MeSH Terms: conditions — Wounds and Injuries; Athletic Injuries; Knee Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes Meeting Return-to-Sport (RTS) Criteria: This group includes athletes who have undergone anterior cruciate ligament reconstruction (ACLR) using a Peroneus Longus tendon graft and meet the return-to-sport (RTS) criteria. These athletes demonstrate psychological readiness, self-reported knee function, and sufficient strength recovery (isokinetic strength at 60°/s, 120°/s, and 240°/s), with an H/Q ratio ≥ 90% and IKDC score ≥ 90. These athletes are eligible to return to their pre-injury sport levels based on the established RTS criteria. They will be assessed for psychological readiness using the ACL-RSI scale, knee function with the IKDC score, and isokinetic strength testing at various velocities.
- Athletes Not Meeting Return-to-Sport (RTS) Criteria: This group includes athletes who have undergone ACLR using a Peroneus Longus tendon graft but do not meet the RTS criteria. These athletes may experience insufficient psychological readiness, self-reported knee function, or muscle strength recovery. Specifically, they may have an H/Q ratio below 90%, an IKDC score lower than 90, or fail to achieve adequate isokinetic strength at the required angular velocities (60°/s, 120°/s, 240°/s). These athletes will be assessed using the ACL-RSI scale, IKDC score, and isokinetic strength testing, and the study will explore the factors contributing to their inability to meet RTS criteria.

SUMMARY:
This clinical trial aims to investigate the correlation between psychological readiness, knee function, and isokinetic performance after anterior cruciate ligament reconstruction (ACLR) using the Peroneus Longus tendon graft (PLT). ACL injuries are common among athletes, and the standard treatment is ACL reconstruction surgery (ACLR). However, the success of the surgery does not solely depend on physical recovery but also on the psychological readiness of athletes to return to their sport.

This study focuses on athletes who have undergone ACLR using the Peroneus Longus tendon (PLT). The primary objective is to compare psychological readiness, self-reported knee function (IKDC score), isokinetic performance (quadriceps and hamstring strength), and muscle strength ratios between athletes who meet return-to-sport (RTS) criteria and those who do not.

Psychological readiness will be assessed using the ACL-Return to Sport after Injury (ACL-RSI) scale, while knee function will be evaluated using the IKDC subjective score. Isokinetic testing will assess quadriceps and hamstring strength at various angular velocities. This study aims to provide a more comprehensive understanding of the factors influencing an athlete's ability to return to sport after ACLR, combining both physical and psychological aspects.

The results will help optimize rehabilitation strategies by offering a multidimensional approach, considering both physical and psychological factors, to improve recovery protocols for ACL-injured athletes.

DETAILED DESCRIPTION:
Rationale and Objectives Anterior cruciate ligament reconstruction (ACLR) using a Peroneus Longus autograft is increasingly adopted; however, return-to-sport (RTS) decisions often emphasize strength or hop metrics while under-weighting psychological readiness. This single-center case-control study evaluates whether athletes who meet a predefined RTS test battery ("RTS-ready") differ from athletes who do not ("RTS-not-ready") in psychological readiness, knee function, isokinetic performance, hamstring-to-quadriceps (H/Q) strength ratio, and dynamic postural control/core endurance. The central hypothesis is that an integrated profile (physical + psychological) characterizes RTS-ready athletes and can inform safer, individualized RTS decisions after ACLR with Peroneus Longus.

Design and Setting Observational, case-control, cross-sectional assessment conducted in a university sports rehabilitation laboratory. Participants attend a single evaluation visit between 6 and 9 months post-ACLR after completing a standardized postoperative rehabilitation pathway. Group assignment (Case = RTS-ready; Control = RTS-not-ready) is determined by performance on the prespecified RTS battery during the same visit.

Participants Key inclusion and exclusion criteria (e.g., male recreational athletes in cutting/jumping sports; primary unilateral ACLR with Peroneus Longus autograft; exclusion of revision/multi-ligament injuries, significant pain or ROM limitation) are listed in the Eligibility Criteria section and are not repeated here.

Procedures and Test Order

All testing is performed in a single session by trained assessors after informed consent and a brief familiarization to minimize learning effects. To standardize workload and reduce fatigue and order effects, assessments proceed as follows:

Self-report instruments: psychological readiness and knee function questionnaires (validated Arabic versions).

Standardized warm-up: 5-10 minutes of low-intensity cycling followed by dynamic lower-limb mobility.

Isokinetic strength testing: HUMAC NORM dynamometer with standardized positioning (seating/strapping), axis alignment to the lateral femoral condyle, and knee range of motion set to approximately 0-90°. After practice trials, peak concentric torque for quadriceps and hamstrings is recorded at 60°/s, 120°/s, and 240°/s per manufacturer guidelines and lab SOPs. Rest intervals of at least 60-90 seconds are provided between sets. Limb Symmetry Index (LSI) is calculated as (involved/uninvolved) × 100 for each parameter. The H/Q ratio is calculated as peak hamstring torque divided by peak quadriceps torque at each speed.

Functional performance tests: single-leg hop for distance (best of three valid trials per limb; hands on hips; controlled landing), Y-Balance Test (anterior, posteromedial, posterolateral reaches normalized to limb length), and prone plank (time to task failure using standardized termination criteria).

Vital signs and knee discomfort are monitored throughout; testing is stopped if predefined safety thresholds are exceeded.

RTS Battery and Group Assignment The RTS battery used for group assignment (e.g., LSI thresholds for isokinetic quadriceps/hamstrings, single-leg hop LSI, and IKDC threshold) is defined in the Outcome Measures section. Participants meeting all criteria are classified as RTS-ready (Case), otherwise RTS-not-ready (Control). Assessors collecting raw measurements remain blinded to RTS labels until all tests are completed and the RTS algorithm is applied.

Quality Control and Bias Minimization The dynamometer undergoes daily calibration verification and periodic full calibration per manufacturer schedule. Scripted instructions and standardized verbal encouragement are used. Equipment setup (seat/backrest angles, lever arm length, strap positions) is recorded to ensure consistency. Any protocol deviations, adverse events, or premature terminations are documented. Data are double-entered and range-checked prior to analysis.

Outcomes Primary and secondary outcomes (psychological readiness, knee function, isokinetic peak torque/LSI, H/Q ratio, hop performance, Y-Balance, and core endurance), including instruments, scoring ranges, directionality, and time frame (single visit at 6-9 months post-op), are fully specified in the Outcome Measures section of this record.

Sample Size and Statistical Analysis A priori sample-size estimation targeted 80% power (two-sided α = 0.05) to detect a moderate between-group effect size in the primary outcomes; detailed parameters are provided in the Statistical Analysis Plan (if uploaded). Data will be screened for normality (e.g., Shapiro-Wilk) and outliers; continuous variables will be summarized as mean ± SD (or median [IQR] if non-normal), categorical variables as counts (%). Between-group comparisons will use independent-samples t-tests (or Mann-Whitney U where assumptions are violated) and chi-square or Fisher's exact tests for categorical variables. Exploratory multivariable logistic regression will estimate the independent association of psychological readiness, strength (LSI), H/Q ratio, and functional tests with RTS status while adjusting for potential confounders (e.g., age, BMI, time since surgery). Effect sizes (Cohen's d or odds ratios with 95% CIs) will be reported. Missing data will be handled with complete-case analysis; if >5% of a primary outcome is missing, sensitivity analyses will be performed. Statistical significance is set at p < 0.05. Analyses will be conducted using SPSS (Version 29.0).

Ethics and Safety The study complies with the Declaration of Helsinki and has Institutional Review Board approval. Written informed consent is obtained before participation. The procedures are non-invasive and considered minimal risk; predefined stop rules are applied for pain or adverse symptoms.

Expected Impact By integrating psychological readiness with objective strength and functional performance, this study aims to refine RTS decision-making after ACLR using Peroneus Longus autografts, potentially reducing re-injury risk and enabling more individualized rehabilitation progressions.

ELIGIBILITY:
Inclusion Criteria:

* Male recreational athletes aged 18-35 years.
* Participation in sports that involve deceleration, jumping, cutting, or turning (e.g., basketball, soccer, volleyball).
* Primary unilateral ACL injury treated with ACL reconstruction using a Peroneus Longus autograft.
* Single evaluation 6-12 months after ACL reconstruction.
* Completed a standardized postoperative rehabilitation program for ≥6 months, with near-complete rehabilitation and some level of sport participation.
* Sufficient knee confidence, no effusion/edema, full knee range of motion, and able to perform all functional tests safely.
* Able to provide written informed consent.

Exclusion Criteria:

* Revision ACL reconstruction.
* Prior ACL reconstruction on the ipsilateral or contralateral knee.
* Multi-ligament knee injury.
* Concomitant meniscal repair or bilateral ACL reconstruction.
* Knee pain > 3/10 at evaluation that prevents or impairs testing.
* Incomplete knee extension or knee flexion < 110°.
* Lower-limb fracture or surgery within the past 6 months.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of male recreational athletes who have undergone anterior cruciate ligament reconstruction using the Peroneus Longus tendon. These athletes must meet specific criteria to return to sport and will be evaluated for both physical and psychological readiness. Participants will be assessed at least 6 months post-surgery, with both case (RTS) and control (non-RTS) groups based on their ability to return to sport.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Psychological Readiness to Return to Sport | Up to 9 months post-operative
  Psychological readiness to return to sport measured by the validated Arabic version of the ACL-Return to Sport after Injury (ACL-RSI). Total score 0-100; higher scores indicate greater psychological readiness.
Isokinetic Strength Performance (Quadriceps Strength at Various Velocities) | Up to 9 months post-operative
  This measure evaluates quadriceps strength at 60°/s, 120°/s, and 240°/s using the HUMAC NORM Isokinetic Dynamometer. It assesses peak torque and average power production in both the injured and uninjured limbs.

SECONDARY OUTCOMES:
Knee Function | Up to 9 months post-operative
  Evaluated using the IKDC subjective score, this measure assesses knee function and symptoms, including limitations in daily and sports-related activities. A higher score indicates better knee function.
Isokinetic Performance (Quadriceps and Hamstring Strength at Different Velocities) | Up to 9 months post-operative
  This outcome measures the strength of quadriceps and hamstrings at 60°/s, 120°/s, and 240°/s. The focus is on measuring peak torque, average power, and Hamstring-to-Quadriceps (H/Q) ratio to assess muscle strength recovery and balance.
Dynamic Postural Control | Up to 9 months post-operative
  This measure evaluates an athlete's dynamic stability and ability to maintain balance through the Y-Balance Test, a functional movement test essential for preventing re-injury.
Core Muscle Endurance | Up to 9 months post-operative
  The Prone Plank Test assesses the endurance of the core muscles, which are vital for overall stability, balance, and functional movements after ACL reconstruction.
Limb Symmetry Index (LSI) | Up to 9 months post-operative
  LSI compares strength between the injured and uninjured limbs. A LSI ≥ 90% is generally considered a benchmark for safe return to sport. It will be calculated based on isokinetic strength testing.
Functional Knee Tests (Single-Leg Hop Test) | Up to 9 months post-operative
  This measure evaluates the ability of the athlete to perform dynamic movements, such as hopping, as part of functional recovery and readiness for return to sport.

CONTACTS AND LOCATIONS:
Locations (1):
- AHUC, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No